CLINICAL TRIAL: NCT02396979
Title: Intervention of HIV, Drug Use and the Criminal Justice System in Malaysia
Acronym: Harapan
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: University of Malaya (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 0908005646; R01DA025943 (NIH)
Record Dates: First submitted 2015-02-23; First posted 2015-03-24 (Estimated); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Human Immunodeficiency Virus; Acquired Immunodeficiency Syndrome; Opiate Addiction; Drug Dependence
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Opioid-Related Disorders; Substance-Related Disorders | interventions — Methadone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Methadone Maintenance (Experimental): Methadone induction and management provided
  Interventions: Drug: Methadone
- Holistic Health Recovery Program (Experimental): Administration of the Holistic Health Recovery Program (HHRP-M), which is an eight-session substance abuse relapse prevention and harm reduction program administered by a trained substance abuse counselor.
  Interventions: Behavioral: Holistic Health Recovery Program
- Methadone Maintenance and Holistic Health Recovery Prorgram (Experimental): Methadone induction and management provided in combination with the Holistic Health Recovery Program (HHRP-M).
  Interventions: Drug: Methadone; Behavioral: Holistic Health Recovery Program
- Standard of Care (No Intervention): Standard of care provided for substance abuse treatment. No methadone maintenance or holistic health recovery program intervention provided.

INTERVENTIONS:
Drug: Methadone
  Arms: Methadone Maintenance; Methadone Maintenance and Holistic Health Recovery Prorgram
Behavioral: Holistic Health Recovery Program
  Arms: Holistic Health Recovery Program; Methadone Maintenance and Holistic Health Recovery Prorgram

SUMMARY:
The purpose of this study is to evaluate the relative impact a medical drug (methadone) or behavioral counseling program (Holistic Health Recovery Program) or both (methadone and Holistic Health Recovery Program) has on reducing HIV-related risk behaviors and illicit drug use among opioid-dependent, HIV-infected individuals in prison when given 90 to 180 days prior to leaving prison.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected
* Clinical Diagnosis of Opioid Dependence
* Fluent in Bahasa Malaysia or English
* Within 90 to 180 days of release from prison
* Planning to live in Klang Valley region after release from prison
* Able to provide informed consent

Exclusion Criteria:

* Pregnancy or planning to become pregnant (female only)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2010-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
HIV Risk Events | Change from Baseline in HIV Risk Events at Months 3, 6, 9 and 12
  The primary outcome is the number of HIV high risk events. This outcome will be constructed from a composite measure counting the number of unprotected vaginal and anal insertive events and needle-or-syringe-sharing events with an HIV- or HIV-status-unknown partner that might result in HIV transmission to an uninfected partner. As such, the primary outcome will be the number of high-risk events during the period of observation in the intervention. All data will be self-reported by the participant.

SECONDARY OUTCOMES:
HIV Quality of Life | Change from Baseline in HIV Quality of Life at Months 3, 6, 9 and 12
  This outcome will be measured by a series of questions that will be used to produce a composite score that will indicate the participant's overall quality of life as it relates to their HIV status. These questions will ask about your general health and your ability to perform daily activities in your life. All data will be self-reported by the participant.
Relapse to Drug Use | Change from Baseline in Relapse to Drug Use at Months 3, 6, 9 and 12
  This outcome will be measured as any opioid drug use after release from prison. This outcome will be measured in two ways. First, participants will provide a monthly urine sample that will be tested for the presence of opioids. Second, participants will answer questions about their drug use since the time of their last interview.
Addiction Severity | Change from Baseline in Addiction Severity at Months 3, 6, 9 and 12
  This outcome will be measured by a series of questions about the participant's drug use. These questions will be used to produce a composite score which indicates the severity of the participant's addiction.
Reincarceration | Any reincarceration to prison during the 12 month post-release follow-up period
  This outcome will be measured by both self-report and objective data from the Malaysian Ministry of Prisons. Self-report questions will be used to ask participants if they have been arrested by police (placed in jail) or incarcerated in prison during the time since the last interview. Objective data will also be obtained from the Ministry of Prisons which will indicate if the participant has been reincarcerated in one of Malaysia's prison during the 12 months since they were initially released from prison.

CONTACTS AND LOCATIONS:
Overall Officials: Frederick L Altice, M.D., Principal Investigator — Yale University; Adeeba Kamarulzaman, M.D., Principal Investigator — University of Malaya

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bazazi AR, Culbert GJ, Wegman MP, Heimer R, Kamarulzaman A, Altice FL. Impact of prerelease methadone on mortality among people with HIV and opioid use disorder after prison release: results from a randomized and participant choice open-label trial in Malaysia. BMC Infect Dis. 2022 Nov 11;22(1):837. doi: 10.1186/s12879-022-07804-6. PMID 36368939
- [Derived] Chandra DK, Bazazi AR, Nahaboo Solim MA, Kamarulzaman A, Altice FL, Culbert GJ. Retention in clinical trials after prison release: results from a clinical trial with incarcerated men with HIV and opioid dependence in Malaysia. HIV Res Clin Pract. 2019 Feb;20(1):12-23. doi: 10.1080/15284336.2019.1603433. Epub 2019 May 1. PMID 31303149